CLINICAL TRIAL: NCT03730974
Title: The Efficacy and Appropriateness of Ball Blankets on Insomnia in Depression in Outpatient Clinics
Brief Title: Ball Blankets on Insomnia in Depression in Outpatient Clinics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Innovation Fund Denmark (Individual); Protac A/S (Unknown); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7777BB
Record Dates: First submitted 2018-07-02; First posted 2018-11-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Insomnia Due to Mental Disorder

STUDY DESIGN:
Intervention Model Description: The study has a randomized 2-sequence, 2-period, 2-treatment crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm AB (Ball blanket + TAU) (Experimental): Participants will be randomized into either sequence AB or BA each lasting four weeks.
  Patients that are randomized to the AB sequence receive intervention A (Protac Ball BlanketTM 7 kg Flexible) in the first two weeks and treatment B treatment as usual (TAU) in the second period.
  Interventions: Device: Protac Ball BlanketTM (7kg Flexible)
- Experimental arm BA (TAU + Ball blanket) (Experimental): Patients that are randomized to the BA sequence receive treatment B (TAU) in the first period and intervention A in the second period (Protac Ball BlanketTM 7kg Flexible).
  Interventions: Device: Protac Ball BlanketTM (7kg Flexible)

INTERVENTIONS:
Device: Protac Ball BlanketTM (7kg Flexible) — All patients will wear a MotionLogger Micro Watch from Ambulatory Monitoring Inc. NY in all four weeks during all 24hours of the day.
  Other Names: MotionLogger Micro Watch from Ambulatory Monitoring Inc. NY

SUMMARY:
The objective of the study is to examine the efficacy of Protac Ball BlanketsTM (PBB) and specifically if the PBB will extend the total sleep time of patients with insomnia due to depression in two psychiatric outpatient clinics at Aarhus University Hospital and Odense University Hospital.

Furthermore, it will be examined whether the PBB will reduce the sleep onset latency, number of awakenings, wake after sleep onset, need for sedatives and hypnotics, the self reported symptoms of depression and anxiety and improve the quality of sleep.

45 patients with depression and insomnia who receive outpatient treatment will be included in this study.

The study is a randomized crossover trial. The data collection period lasts four weeks. Data will be collected using actigraphy, sleep diaries and questionnaires.

DETAILED DESCRIPTION:
This PhD project is an industrial PhD. The protocol is approved and fully financed by the Innovation Fund Denmark (case number 7038-00157B), Protac A/S, Skanderborg and Aarhus University, Denmark.

The project will take place at The Mood Disorders Clinic, Aarhus University Hospital, Risskov, Central Denmark Region and in The Clinic of Affective Disorders, Department of Psychiatry, Psychiatry in The Region of Southern Denmark.

Background: Depression affects approximately 5% of the Danish population and is associated with significant morbidity and mortality. Proper treatment of these patients is therefore, an important clinical and public health issue. Unfortunately, some symptoms of depression are difficult to manage which is the case for sleep disturbances such as insomnia. Insomnia occurs in the majority of patients with depression, and is characterized as problems with initiating sleep, several awakenings, early wake ups, poor sleep quality, and daytime dysfunction. The causality of the insomnia-depression relationship is debated. Several studies have raised the question whether insomnia is not just a typical symptom of depression but rather an independent clinical predictor of depression, which implicates the importance for primary prevention and specific focus on the treatment of insomnia. Often, medication is used to treat insomnia but pharmacological treatment has side effects and, importantly, there is a risk of drug tolerance and addiction. Increased attention on investigating the known and un-known benefits of non-pharmacological treatment options for sleep disturbances is therefore highly relevant. Non-pharmacological treatments include cognitive behavioural therapy, which has proven effects on insomnia. Cognitive behavioural therapy for insomnia (CBTI) typically includes sleep restriction, stimulus control, cognitive therapy, sleep hygiene and relaxation training. It has been included as the treatment of choice in a campaign by the Danish National Board of Health. Unfortunately, CBTI is limited to patients without severe cognitive problems that are mentally able to participate in therapy sessions. Therefore, more evidence based non-pharmacological treatment options that hit a greater target group are needed if tailor-made management of insomnia in depression is to be achieved.

Ball blankets are a promising option that can be used in all patients including patients with severe cognitive deficits due to depression. It has been shown to decrease sleep disturbances in children with ADHD using the Protac Ball BlanketTM (Protac A/S, Skanderborg, Denmark). The Protac Ball BlanketTM (PBB) has been used in adult psychiatric inpatient settings since the early 1990s for patients suffering from insomnia, anxiety, agitation, manic episodes and psychosis. From a clinical perspective the blankets is experienced to enhance the patient's awareness of the body and its physical delimitation which relieves restlessness, stress and anxiety and provides a sense of security and calm in head and body, which for some resolves in improved sleep quality. This is in line with the mechanism of the PBB, which is to provide a changing sensory stimulation because of the movement of the plastic balls in the blanket. Further, the weighted plastic balls gives a light pressure distributed across numerous points, helping the brain to register the body. During sleep the balls will move because of slight changes in body position and the skin is thus continuously stimulated in new ways.

Clinical experiences support the use of PBB in depression but there are neither RCTs nor qualitative studies on the effects and appropriateness of using PBB in insomnia among adults with depression. Two dissertations on sleeping problems due to dementia or sense of touch and sense of movement issues in kids indicate effects of using ball blankets. Overlap in symptoms between these conditions and depression, i.e. anxiety and sleep disturbances suggests an effect in depression. Currently, ball blankets are used as an unapproved treatment option among adults with depression. However, lack of solid evidence limits the use of PBB in the adult population or may expose some to a useless treatment. Further, if ball blankets are beneficial for a proportion of patients with depression, the lack of data on adult patient hampers further development and improvement of the PBB for the benefit of patients.

Possible reasons for insomnia in depression are: anxiety, stress, agitation and suicidal thoughts. Additional, insomnia plays a role in several biological processes such as stress and mood regulations, therefore an important goal in the treatment of depression is to normalize the total sleep time, minimize the sleep onset latency and improve quality of sleep, and at the same time minimize the use of sedatives. Investigators hypothesize that PBB will extend sleep durations, minimize the sleep onset latency, reduce the number of awakenings, reduce the need for sedatives, improve the quality of sleep and reduce the self-reported symptoms in patients with insomnia due to depression.

Since 2007 the duration of inpatient treatment has been shortened significantly. Consequently, fewer patients with depression are in remission at hospital discharge. Importantly, some will still be weeks from the full effect of the antidepressant medication when discharged as the full pharmacological treatment may take from 6-8 weeks to reach and an average hospital admission is estimated to 19 days. Therefore many patients still suffer from fatigue due to the disturbances in sleep associated with depression. Medical treatment for sleep disorders may be problematic as described. The fatigue in itself makes coping with everyday life challenging and hinders the rehabilitation process.

Furthermore, depression-related financial costs in Europe are estimated at €113,4 billion every year due to health care costs and reduced ability to work. From a financial perspective, this illustrates the importance of reducing the symptoms and duration of the depressions (and this is of cause obvious from an individual and clinical perspective). If the non-pharmacological treatment with PBB has an effect it may thus potentially reduce social-, health- and socio-economic costs because of the reduced fatigue in important stages of depression and potentially faster return to normality for the patients.

PBB is potentially an innovative non-pharmacological alternative to the medical treatment of patients with insomnia due to depression but solid evidence is needed, before the treatment can be implemented. Furthermore clinical data from this project may improve the product.

Objective: To investigate the efficacy of PBB on insomnia in adult patients with depression in outpatient psychiatric clinics.

Hypotheses: The use of PBB on patients with insomnia due to depression will:

Primary goal:

1. Extend the total sleep time

Secondary goals:

1. Reduce sleep onset latency
2. Reduce the number of awakenings
3. Reduce wake after sleep onset
4. Reduce the need for sedatives and hypnotics
5. Improve the quality of sleep
6. Reduce the self-reported symptoms of patients with depression

Methods: The study is carried out as a randomized crossover trial. The study has a randomized 2-sequence, 2-period, 2-treatment crossover design.

Sample size: The power calculation is based on a literature review and a pilot study (N=8). The main outcome will be changes in total duration of sleep. The null hypothesis is no change in sleep duration. In the pilot study, the mean sleep duration was 420 minutes. The standard deviation of the difference within each person was 42 minutes. It is a cross-over design and investigators will perform a paired, two-sided analysis. The aim is to be able to detect a change in total sleep time of 20 minutes and with an alfa=0.05 and beta=0.20 the minimum sample size based on the pilot study is N=37. To take into account drop out rates investigators aim to include 45 patients.

Variables and Assessment: The total sleep time, sleep onset latency, number of awakenings and wake after sleep onset will be assessed by actigraphy (MotionLogger Micro Watch from Ambulatory Monitoring Inc. NY) and sleep diaries including "bed time" and "time getting out of bed" registrations. The severity of depression and anxiety will be assessed using 6-item Hamilton Rating Scale for Depression (HRSD6), the Major Depression Inventory (MDI), Self Reported Symptoms (SCL-28) and Becks Anxiety Index (BAI). The severity of Insomnia will be assessed using the Insomnia Severity Index (ISI) and Sleep quality will be assessed using the Pittsburg Sleep Quality Index (PSQI).

Data analysis Data will be analyzed using MotionLogger Analysis Software Programs (from Ambulatory Monitoring Inc. NY) and Stata 15 (StataCorp, Tx, USA). The computer generated randomization will determine whether the participants will begin or end with a weight blanket. The baseline characteristics of these two groups will be presented in a table to illustrate the result of the randomization. The "ladder" command in Stata will be used to search for potential transforms that convert the continuous outcome measures into normally distributed variables, and the measures will be transformed accordingly. For the scores, e.g. PSQI, the study will estimate changes in the score and therefore the measures are likely to be normally distributed even though the underlying score is not. If normality is impossible to reach for some measures, even after transformation, non-parametric tests will be used, e.g. Wilcoxon signed-rank tests or Fisher's exact tests. An intention to treat analysis will be conducted and the outcome measures (potentially transformed) will be compared using a paired sample t-test. The level of statistical significance will be set to 5%.

ELIGIBILITY:
Inclusion Criteria:

* Participants: Patients with depression according to ICD-10 (F32-33) or (F32-33 in combination with F40-41.2) (males and females, aged ≥18 years) who receive outpatient treatment in The Mood Disorders Clinic, Aarhus University Hospital, Risskov, Denmark and in The Clinic of Affective Disorders, Department of Psychiatry, Psychiatry in The Region of Southern Denmark.
* Participants must either experience poor sleep quality, sleep onset latency or wake time after sleep onset of: (a) ≥31 min; (b) occurring ≥3 nights a week; (c) for ≥ 14 days (31) or early wake ups, and have a Global Pittsburgh Sleep Quality Index Score ≥5.

Exclusion Criteria:

* Patients that, according to ICD-10 criteria, have been depressed >2 years
* Patients suffering from hypersomnia (ICD-10: F51.13)
* Patients with current alcohol- or drug abuse (ICD-10: F10-19)
* Patients with diseases directly influencing sleep quality (such as severe chronic pain issues, sleep apnoea o.a.)
* Patients receiving medications causing sleep loss and disturbed sleep
* Patients with Circadian Rhythm Sleep-Wake Disorders (ICD-10; G47.20-47.26)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in total night time sleep (TST) measured by actigraphy (Micro MotionLogger Watch) | Four weeks
  The investigators will detect the change in total night time sleep in minutes (actual sleep time, excluding sleep latency and wakes after sleep onset) by comparing the means of the difference in TST for each participant between period A and B or B and A

SECONDARY OUTCOMES:
Changes in sleep onset latency (SOL) | Four weeks
  The investigators will measure patients' SOL in minutes (time between registered bed time in sleep diaries and first sleep onset measured by actigraphy) and compare the means of the difference for each participant between periods
Changes in number of awakenings measured by actigraphy (Micro MotionLogger Watch) | Four weeks
  The investigators will measure the number of awakenings between first sleep onset and the last wake up time registry and compare the means of the difference between period A and B or B and A for each participant
Sedatives and hypnotics measured by medication registration use in sleep diaries | Four weeks
  The investigators will measure the change in use of per need sedatives and hypnotics in mg by comparing the means of the difference for each participant between periods
Quality of sleep measured by questionnaire using the Pittsburgh Sleep Quality Index | Data will be collected at baseline, after two weeks and after four weeks. The difference between PSQI measured at week 2 and week 0 will be compared with the difference in PSQI measured at week 4 and week 2.
  The investigators will measure and report the change in quality of sleep between periods. The total Pittsburgh Sleep Quality Index Score between 0-21, where "0" indicating no difficulty and "21" indicating severe difficulties is reported.
Symptoms of depression measured by the self-reported Hamilton Depression Rating Scale (HRSD6) | Data will be collected at baseline, after two weeks and after four weeks. The difference between the score measured at week 2 and week 0 will be compared with the difference in score measured at week 4 and week 2.
  The investigators will measure the change in self-reported symptoms of depression between periods. The total sum score between 0-50 is reported, where higher values represent worse outcome
Insomnia Severity Status measured by questionnaire using the Insomnia Severity Index | Data will be collected at baseline, after two weeks and after four weeks. The difference between the score measured at week 2 and week 0 will be compared with the difference in score measured at week 4 and week 2.
  The investigators will measure the change in patients' insomnia severity status. The total score between 0-28 is reported, where higher values represent worse outcome
Patients self-reported symptoms of depression measured by questionnaire using Major Depression Inventory (MDI) | Data will be collected at baseline, after two weeks and after four weeks.The difference between the score measured at week 2 and week 0 will be compared with the difference in score measured at week 4 and week 2.
  The investigators will measure the change in self-reported symptoms of depression between periods. The total score between 0-50 is reported, where higher values represent worse outcome.
Symptoms of anxiety measured by questionnaire using Beck Anxiety Index (BAI) | Data will be collected at baseline, after two weeks and after four weeks.The difference between the score measured at week 2 and week 0 will be compared with the difference in score measured at week 4 and week 2.
  The investigators will measure the change in self-reported symptoms of anxiety between periods. The total score between 0-63 is reported, where higher values represent worse outcome.
Patient-reported outcomes concerning interpersonal sensitivity, neurasthenia, anxiety, and depression measured by questionnaire using The Self-Reported Symptom State Scale SCL-28 | Data will be collected at baseline, after two weeks and after four weeks.The difference between the score measured at week 2 and week 0 will be compared with the difference in score measured at week 4 and week 2.
  The investigators will measure the change in self-reported symptoms between periods. Sub scales are combined to compute a total score. The range for each sub scale are: Interpersonal Sensitivity 0-32, Neurasthenia 0-28, Anxiety 0-32 and Depression 0-24. Both total score and sub scale scores will be reported. The total score range between 0-112, where higher value represent worse outcome. Because of an overlap in one question between the sub scales anxiety and depression question number 31 is only considered in the total sum ones.
Changes in wake after sleep onset (WASO) measured by actigraphy | Four weeks
  The investigators will measure patients total time awake between initial sleep onset and the final morning awakening in minutes and compare the means of the difference between period A and B or B and A for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Erik R Larsen, MD PhD, Study Director — Odense University Hospital
Locations (2):
- Denmark (2):
  - The Mood Disorders Clinic, Aarhus, Central Danish Region
  - Mental Health Department Odense - University Clinic, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristiansen ST, Videbech P, Bjerrum MB, Larsen ER. The efficacy of ball blankets on insomnia in depression in outpatient clinics: study protocol for a randomized crossover multicentre trial. Trials. 2020 Aug 17;21(1):720. doi: 10.1186/s13063-020-04638-y. PMID 32807208